CLINICAL TRIAL: NCT03190720
Title: Development of Exercise Promotion Program Using a Mobile Community Based on a Smart Phone Application in Breast Cancer Survivors
Brief Title: Development of Exercise Promotion Program Using a Mobile Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Il Yong Chung, Clinical Assistant Professor, Asan Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-0328
Record Dates: First submitted 2017-06-12; First posted 2017-06-19 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer; Physical Activity
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: two different single-arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Community First (Experimental): Participants will be registered to a mobile community at first. After 6 weeks, They will leave the mobile community.
  Interventions: Device: Mobile community
- Mobile Community Later (Experimental): Participants will not be registered to a mobile community at first. After 6 weeks, They will be registered to the mobile community.
  Interventions: Device: Mobile community

INTERVENTIONS:
Device: Mobile community — A mobile community based on smartphone application (WalkOn) which gives participants to information about their own steps and others'.

SUMMARY:
This study aims to investigate the effect of a mobile community based on a smart phone application to enhance physical activities of breast cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Stage 0-III breast cancer

Exclusion Criteria:

* Stage IV breast cancer
* Breast cancer recurrence or metastasis
* Severe medical illness

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Distress | up to 3months
  Assessment using Patient Health Questionnaire (PHQ-9)

SECONDARY OUTCOMES:
Physical activity | up to 3months
  Assessment using International Physical Activity Questionnaire (IPAQ)

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Korea, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chung IY, Jung M, Park YR, Cho D, Chung H, Min YH, Park HJ, Lee M, Lee SB, Chung S, Son BH, Ahn SH, Lee JW. Exercise Promotion and Distress Reduction Using a Mobile App-Based Community in Breast Cancer Survivors. Front Oncol. 2020 Jan 10;9:1505. doi: 10.3389/fonc.2019.01505. eCollection 2019. PMID 31998651